CLINICAL TRIAL: NCT03197272
Title: Non-invasive Phototherapeutic Intrastromal Corneal Collagen Crosslinking (PiXL) for Low-grade Myopia
Brief Title: Advanced Cross Linking for Low-grade Myopia
Acronym: PiXLO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PiXLMYOP-I
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Myopia; Corneal Crosslinking
Keywords: Myopia; corneal Crosslinking
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Prospective, single-masked intraindividually comparing randomized controlled trial. Participants will be randomized to receive ultraviolet (UV) light according to protocol A in one eye and protocol B in the other, which is masked to the participant. Both eyes will be treated during the same visit.
  Protocol A: UV irradiation in a central 4 mm homogenous zone of the cornea. Protocol B: UV irradiation in a central ring-shaped 4 mm area of the cornea. Patients are randomized utilizing a computer list of unique random numbers between 1 and 23; an even number will be treated with a homogeneous zone in the right eye; an uneven number with a homogeneous zone in the left eye.
Who Masked: Participant
Masking Description: The participants are not aware which eye will receive the homogeneous zone treatment and which eye will receive the ring-shaped treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PiXL Protocol A (Experimental): PiXL treatment with UV irradiation in a central 4 mm homogenous zone of the cornea. For myopia of less than 1.0D, 10 J/cm2 will be used, for higher levels of myopia 15J/cm2 will be used.
  Interventions: Procedure: PiXL
- PiXL Protocol B (Active Comparator): PiXL treatment with UV irradiation in a central ring-shaped 4-mm area of the cornea. A central 2-mm zone is left untreated, and the energy is higher towards the periphery of the ring-shaped area, reaching its maximum at 2 mm from the corneal centre. For myopia of less than 1.0D, a maximum of 10 J/cm2 will be used, for higher levels of myopia a maximum of 15J/cm2 will be used.
  Interventions: Procedure: PiXL

INTERVENTIONS:
Procedure: PiXL — Phototherapeutic intrastromal corneal collagen cross-linking (PiXL) performed in a high-oxygen environment without corneal epithelial debridement, for treatment of mild myopia.

SUMMARY:
To evaluate the improvement in myopic refractive error and the corneal endothelial safety with a corneal crosslinking treatment regimen for mild myopia. The treatment involves a 4-mm central treatment zone in high oxygen environment without corneal epithelial debridement.

DETAILED DESCRIPTION:
The study is designed as a prospective, single-masked intraindividually comparing randomized controlled trial involving healthy volunteers ≥18 years of age of both genders with mild myopia, performed at the Department of Clinical Sciences / Ophthalmology, Umeå University Hospital, Umeå, Sweden. The study involves 23 persons with a myopia of -0.5 to -2.5 diopters (D) and astigmatism of ≤0.75 D. All participants are treated with phototherapeutic intrastromal corneal collagen cross-linking (PiXL) without epithelial debridement (epi-on), after topical riboflavin. For myopia of less than 1.0D, 10 J/cm2 will be used, for higher levels of myopia 15J/cm2 will be used, and the treatment involves continuous delivery of oxygen around the eye using an oxygen mask to achieve an oxygen concentration of ≥90% during treatment. Participants will be randomized to receive ultraviolet (UV) light according to PiXL Protocol A in one eye and PiXL Protocol B in the other, which is masked to the participant. Both eyes will be treated during the same visit.

Protocol A: UV irradiation in a central 4 mm homogenous zone of the cornea. Protocol B: UV irradiation in a central ring-shaped 4 mm area of the cornea. Patients are randomized utilizing a computer list of unique random numbers between 1 and 23; an even number will be treated with a homogeneous zone in the right eye; an uneven number with a homogeneous zone in the left eye. All patients are informed about the procedures and provide oral and written consent before inclusion in the study.

At baseline, before treatment, each eye is evaluated with slit-lamp examination, subjective refraction, determination of uncorrected (UCVA) and best corrected (BSCVA) visual acuities using the LogMAR fast protocol and intraocular pressure (IOP) using Goldmann applanation tonometry. Each eye is photographed using the "25 pictures" program with the Pentacam HR® (Oculus, Inc. Lynnwood, WA) under standardized, mesopic light conditions. Keratometry readings, central corneal thickness and the average corneal densitometry values (corneal light backscatter), expressed as standardized gray scale units, GSU) is determined with the Pentacam HR®. Central corneal endothelial photographs are taken with the Topcon SP-2000P specular microscope (Topcon Europe B.V., Capelle a/d Ijssel, the Netherlands), and the corneal endothelial cell count is calculated from a cluster of 25 cells from each photograph.

All the above mentioned investigations are repeated at 1, 3, 6,12 and 24 months after the treatment. At 1 week after treatment, UCVA is registered and a slit-lamp examination, a subjective comparison of discomfort and visual performance in each eye and an autorefractometer measurement are performed. One day after treatment the latter 3 examinations are performed.

ELIGIBILITY:
Inclusion Criteria:

* Spherical equivalent on distance subjective refraction between -0.50D and -2.50D.
* Astigmatism ≤ 0.75D
* Stable myopia. Maximum change in refraction of 0.50D in the last 2 years.
* Best corrected visual acuity of at least 0.00 logMAR (ETDRS chart).
* Thinnest pachymetry reading ≥ 440 μm.
* No previous ocular surgery.
* No cognitive insufficiency interfering with the informed consent.

Exclusion Criteria:

* History of or current ocular condition, disease, surgery or medication with ocular effects that could affect the outcomes of the treatment.
* Allergy to any substance or device used in the study.
* Cognitive insufficiency interfering with the informed consent.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in uncorrected visual acuity | 1, 3, 6 and 12 months after treatment
  Change from baseline in distance uncorrected visual acuity
Change from baseline in spherical equivalent | 1, 3, 6 and 12 months after treatment
  Change from baseline in spherical equivalent on subjective distance refraction

SECONDARY OUTCOMES:
Change from baseline in corneal endothelial cell density | 12 months after treatment
  Change from baseline in central corneal endothelial cell density

CONTACTS AND LOCATIONS:
Overall Officials: Anders Behndig, MD, PhD, Principal Investigator — Department of Clinical Sciences/Ophthalmology, Umeå University, Umeå, Sweden
Locations (1):
- Department of Clinical Sciences/Ophthalmology, Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No